CLINICAL TRIAL: NCT07295834
Title: A Multi-centre, Double-blind Randomised Controlled Trial to Compare Modafinil Versus Placebo Over 12 Weeks in Patients With Severe Fatigue and Inflammatory Bowel Disease (MFI): a Feasibility Study
Brief Title: Modafinil For Fatigue in IBD: A Feasibility Randomised Controlled Trial
Acronym: MFI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 344329; M-2024-2 Moulton (Other Grant/Funding Number: Crohn's and Colitis UK); Jon Moulton Charity Trust (Other Grant/Funding Number: Jon Moulton Charity Trust)
Record Dates: First submitted 2025-11-20; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); Fatigue
Keywords: Crohn's Disease; Fatigue; Ulcerative Colitis; Modafinil
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 1 capsule, increasing if needed after 2 weeks to 2 capsules, increasing if needed after 2 weeks to 3 capsules. Total treatment duration 12 weeks.
  Interventions: Drug: Placebo
- Modafinil (Active Comparator): 1 x 100mg, increasing if needed after 2 weeks to 2 x 100mg, increasing if needed after 2 weeks to 3 x 100mg. Total treatment duration 12 weeks.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — 100-300mg daily according to patient response
  Arms: Modafinil
Drug: Placebo — 1-3 placebo capsules according to patient response
  Arms: Placebo

SUMMARY:
Fatigue is a big problem in people with inflammatory bowel disease (IBD). Even when IBD is well controlled, 50% of patients remain fatigued most of the time. Fatigue can be physical (e.g. feeling tired or weak) and mental (e.g. brain fog). However, there are no effective treatments for IBD fatigue.

Modafinil is a medication that can rapidly improve fatigue. It usually acts within 30 minutes and improves wakefulness. It can also improve brain fog. Modafinil has been used for over 30 years in people with narcolepsy, which is a condition where people fall asleep during the day. Modafinil has also been used in people who do not have narcolepsy.

This study will compare modafinil with a dummy tablet (placebo) in people with IBD. This is a feasibility study. This means it primarily aims to test whether a trial like this can be conducted in people with IBD.

Half of the patients in the study will receive modafinil and half will receive placebo. Treatment will be 12 weeks. Patients will start by taking 1 tablet and will then increase to 2 tablets and then 3 tablets if needed. A computer will randomly allocate treatment, meaning there is an equal chance of being allocated modafinil or placebo. They will be followed up after 6 weeks and 12 weeks.

Being a feasibility study, the investigators will measure how many patients consent to the study; how many complete treatment; and how acceptable the treatment is. Participants will complete a range of questionnaires measuring fatigue, mental health and gut health, primarily to look at the completeness and spread of data, and to obtain estimates of treatment effects and their variance.

If feasible, this study will support a larger version of the trial.

DETAILED DESCRIPTION:
Design: The current study is a randomised controlled trial (a study in which people are allocated by chance to receive different interventions). The trial will compare mirtazapine against a placebo (dummy) tablet in 70 patients with both severe fatigue and IBD. This is a feasibility study, meaning that it is testing whether it will be possible to do a larger version of this study.

Setting: Consent and assessments will take placebo in clinic rooms or clinical research facilities at Imperial College Healthcare National Health Service (NHS) Foundation Trust, King's College Hospital, St Mark's Hospital and Guy's and St Thomas' Hospital, or online if the patient prefers this. The latter is important in maximising participation to the study for participants who may find it difficult to access hospitals, which is a common problem in inflammatory bowel disease (IBD) due to issues like pain and incontinence.

Recruitment: Consecutive patients aged ≥18 with diagnosed IBD and significant fatigue will be identified from outpatient clinics and biologics infusion suites. If possible, clinicians will use the IBD Fatigue Scale to identify people scoring ≥11. If necessary, patients will be identified from screening of endoscopy schedules and IBD multidisciplinary team meetings. The clinical team will seek the patient's permission to be contacted by the research team.

If they agree, the research team will then contact the patient - either in the clinic or over the phone - and provide the patient information sheet. The research team will check some basic pre-screening questions: confirming IBD diagnosis, duration of fatigue, whether they are planned to change any IBD treatments in the next 12 weeks, and the 5- question IBD Fatigue Assessment Scale if not already completed. Before pre-screening, the research team will advise patients that the fatigue information they provide will be passed onto their clinical team - with their permission - even if they decide not to take part in the study. They will be advised that any other information about their IBD will not be retained by the study team if they do not wish to take part. If anyone has an elevated fatigue score but does not wish to take part in the study, the research team will seek the patient's permission to relay the fatigue score to their clinical team.

Those who are deemed to be potentially eligible after pre-screening will be invited for a full screening assessment with a member of the study team. Final study inclusion and consent will be taken by a study doctor.

Study procedures: There will be 4 main study visits. At the first visit, the researcher will explain the study in detail. They will answer any questions the participant has. They will ask the participant some brief questions about their mental health and gut health. They will complete the IBD Fatigue Scale if not already done to ensure they score ≥11/20. The research team will confirm that their fatigue is at least 6 months in duration. If eligible according to screening criteria, the research team will invite them to participate and to sign a consent form.

The researchers will check that the participant meets all the inclusion criteria and none of the exclusion criteria. They will ask the participant more detailed questions about fatigue and mental health (the National Institute for Health and Care Excellent (NICE) criteria for chronic fatigue syndrome, Mini Neuropsychiatric Interview for depression) and will complete further questionnaires lasting around 20 minutes. They will also be asked to have height and weight measured and to provide a blood sample (though these are not compulsory). They will have their hand grip strength tested. If female and of childbearing age, the researcher will take a blood pregnancy test. If they are eligible to take part, the participant will then be randomised by computer to one of the 2 treatments (modafinil or placebo). The tablets for both groups are made to look the same. Neither participant nor the research team will know in which treatment group they are allocated to.

Participants will be given medication the same day or will receive it via recorded post.

The 2 treatment arms are:

1. Modafinil (a stimulant medication) If randomised to this group, the participant will be asked to take a modafinil capsule once in the morning. If their fatigue does not improve much, they can add a second tablet after 2 weeks. If needed, they can then add a third tablet after 4 weeks. The total treatment lasts 12 weeks.
2. Placebo If randomised to this group, the participant will take a placebo tablet once per day for 12 weeks. If their fatigue does not improve much, they can add a second tablet after 2 weeks. If needed, they can then add a third tablet after 4 weeks. The total treatment lasts 12 weeks. Participants will not know which treatment (modafinil or placebo) they are taking.

The participant will meet with the research team again at 6 and 12 weeks after starting treatment. This can be in person or online. These appointments will last for around 30 minutes and will involve:

* Repeating most of the questionnaires completed at the beginning
* A review of general health and other medications
* Repeat blood tests and weight measurement (12 weeks only)
* Repeat hand grip strength measurement (12 weeks only)

Although they will finish treatment after 12 weeks, the investigators will participants whether they can attend a final visit 6 weeks later. This is not compulsory. It will involve repeating most of the questionnaires. Throughout, participants will still be able to access any talking therapies for depression or fatigue, though should not start any other antidepressants.

Progression criteria: The milestones for progression to a full efficacy clinical trial will be based on the proportion-to-target of patients randomised overall; % completing 12 weeks of treatment; % of participants taking at least 75% of prescribed mediation; % of planned data and samples collected at 12 weeks; and % participants describing the treatment as acceptable (≥6/10 on 0-10 scale).

Sample size: As a feasibility study, power calculations for a treatment effect are not applicable. The investigators will recruit 70 participants (35 per group), which is sufficient to generate robust variance estimates. Based on 70 patients and an anticipated follow-up rate of 80%, a two-sided confidence interval will extend no more than 12% of the observed proportion.

Data management:

Data will be collected on paper case report form (CRF) and then transferred to an electronic case report form (eCRF). The type of activity that an individual user may undertake is regulated by the privileges associated with his/her user identification code and password. All forms and tapes related to study data will be kept in locked cabinets. Access to the study data will be restricted. The database will be password-protected.

Statistical methods:

A statistical analysis plan (SAP) will be approved by the Trial Steering Committee independent statistician. The analysis population will use intention-to-treat principles. A recruitment plot of predicted vs. actual recruitment will be generated on a monthly basis.

Participant flow through the study will be presented. Descriptive data will be presented in the form of means and standard deviations; medians and ranges; or percentages with 95% confidence intervals, as appropriate depending on the data being described. The investigators will use linear mixed models to estimate the between group adjusted mean difference (aMD) between mirtazapine and placebo groups at week 12 after adjustment for baseline scores, time, and a treatment-by-time-interaction. Associated 95% confidence intervals will be presented alongside the aMD without p-values. More details will be provided in the statistical analysis plan.

Timeline: This 24-month study includes up to 5 months for setup and approval, 12 months for recruitment (plus 3 months' contingency), 4 months for follow-up visits (including post-treatment follow-ups) and 3 months for write-up and dissemination.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of Crohn's disease (CD) or ulcerative colitis (UC) according to clinical notes
2. Reported fatigue duration of 6 months or more
3. Aged 18 years or over
4. Current IBD Fatigue Assessment Scale score ≥11/20
5. Use of contraception if female and of childbearing age. Female participants of childbearing age will require a negative serum/urine pregnancy test before starting the study and will also need to agree to use an acceptable form of contraception throughout the intervention period, e.g. long-acting reversible contraceptive.
6. Faecal calprotectin <250mcg within the last 3 months
7. Normal haemoglobin concentration (≥130g/L [men] and ≥120g/L [women]) within the last 3 months
8. Thyroid stimulating hormone (TSH) level (0.4-4.0 mU/L) within last 3 months
9. Serum total B12 concentration (≥180 nanograms/L) within last 3 months
10. Able to provide written informed consent to enter the trial.

Exclusion Criteria:

1. Diagnosis of drug or alcohol dependence syndrome according to patient report or GP record.
2. Diagnosis of any dementia according to patient report or GP record.
3. Diagnosis of psychosis or schizophrenia according to patient report or GP record.
4. Diagnosis of bipolar disorder according to patient report or GP record.
5. Current active suicidal ideation on clinical assessment by study psychiatrist.
6. Current treatment with stimulant medication (e.g. methylphenidate), dopamine agonist (e.g. ropinirole), levo-dopa (L-DOPA), antipsychotic (e.g. olanzapine), avacopan, avaritinib, bosutinib, doravirine, grazoprevir, leniosilib, moboceritinib, Osimertinib, sofosbuvir, velpatasvir or voxilapravir
7. Contraindications to the administration of modafinil, as per the current SmPC.
8. Patient-reported hypersensitivity to modafinil
9. Non-registration with a GP or failure to consent to sharing of the GP summary care record and any psychiatric assessments held.
10. Currently enrolled in another drug trial or psychological therapy trial.
11. Currently hospitalised for the treatment of IBD.
12. Currently being prescribed a course of budesonide or reducing course of prednisolone for IBD.
13. Planned change in IBD treatment within the next 12 weeks.
14. Currently breastfeeding, pregnant or planning pregnancy.
15. Diagnosis of indeterminate colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 years
  Participants randomised overall, percentage of target
Trial adherence | 12 weeks
  Percentage of participants completing 12 weeks of treatment
Treatment adherence | 12 weeks
  Percentage of participants taking at least 75% of prescribed mediation
Study procedures acceptability and compliance | 12 weeks
  Percentage of planned data and samples collected at primary endpoint (12 weeks)
Overall acceptability | 12 weeks
  Percentage of participants describing the treatment as acceptable (≥6/10 on 0-10 scale)

SECONDARY OUTCOMES:
First 5 questions of the Inflammatory Bowel Disease-Fatigue questionnaire | 12 weeks
  Range 0-20, higher scores indicate worse fatigue
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale | 12 weeks
  Range 0-52, higher scores indicate less fatigue
Patient Health Questionnaire-9 | 12 weeks
  Range 0-27, higher scores indicate worse depression
Generalised Anxiety Disorder-7 | 12 weeks
  Range 0-21, higher scores indicate worse anxiety
Maudsley 3-item Visual Analogue Scale | 12 weeks
  Range 0-300, higher scores indicate worse depression
Pittsburgh Sleep Quality Index | 12 weeks
  Range 0-21, higher scores indicate worse sleep
Euroqol 5-dimension quality of life questionnaire (EQ-5D-5L) | 12 weeks
  Range 0-1, higher scores indicate better quality of life
Harvey Bradshaw Index (Crohn's disease patients only) | 12 weeks
  Higher scores indicate worse disease activity
Simple Clinical Colitis Activity Index (ulcerative colitis patients only) | 12 weeks
  Higher scores indicate worse disease activity
Inflammatory Bowel Disease Control Questionnaire | 12 weeks
  Range 0-16, higher scores indicate better disease activity
Hand grip strength | 12 weeks
  Range 0-100kg, higher scores indicate better hand grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Calum Moulton, Principal Investigator — Imperial College London
Locations (4):
- United Kingdom (4):
  - Imperial College Healthcare NHS Trust, London
  - St Mark's Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT07295834/Prot_SAP_000.pdf